CLINICAL TRIAL: NCT02380781
Title: Contraceptive Counseling in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11-14-40
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Contraceptive Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients will receive current standard postpartum contraceptive counseling.
- Intervention (Experimental): Patients will receive current standard postpartum contraceptive counseling and will be shown a 10 minute video from the CHOICE project which outlines the different contraceptive options
  Interventions: Behavioral: Information in the form of a video

INTERVENTIONS:
Behavioral: Information in the form of a video — see intervention description
  Arms: Intervention

SUMMARY:
This is a prospective randomized control trial in which we propose an intervention in the immediate post-partum period to educate women about contraceptive options, particularly long acting reversible contraception (LARC) methods with an aim of increasing the amount of women who choose a LARC method.

DETAILED DESCRIPTION:
Eligible participants will be identified in the post-partum period and will be randomized to one of two groups. The control group will receive the standard of care contraceptive counseling which includes any prenatal counseling they received as well as information from the nurse practitioner that rounds on them in the post-partum period. The intervention group will also receive the standard of care contraceptive counseling but will also watch a 10 minute video created by the CHOICE project which counsels on different contraceptive options. Both groups will fill out a pre-intervention questionnaire as well as a post-intervention questionnaire 24hrs later. The primary outcome will be which type of contraception each woman chooses. The secondary outcomes will include determining if the women come to their post-partum visits as well as if they get the method of contraception they chose on the post-partum floor.

ELIGIBILITY:
Inclusion Criteria:

* Women giving birth at University Hospitals Case Medical Center
* Patient of the Women's Health Center
* Women delivering only one child
* Women receiving contraceptive counseling from the nurse practitioner that cares for the postpartum unit

Exclusion Criteria:

* Severe neonatal complication at time of delivery (neonatal death, neonatal admission to the neonatal intensive care unit (NICU) except in cases of chorioamnionitis)
* Severe maternal complication at time of delivery (patient requiring intensive care unit care, patient requiring hysterectomy at time of delivery)
* Preterm delivery <34 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Choice of contraceptive method | 24 hours post-intervention
  Will be obtained through use of a questionnaire.

SECONDARY OUTCOMES:
Return to clinic for postpartum visit | 12 weeks post-intervention
  Will use ambulatory electronic medical record (EMR) to determine if patient returned to clinic for follow up visit.
Obtained desired method of contraception | 12 weeks post-intervention
  Will use ambulatory EMR to determine if patient received her desired method of contraception.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer LB, Zolna MR. Unintended pregnancy in the United States: incidence and disparities, 2006. Contraception. 2011 Nov;84(5):478-85. doi: 10.1016/j.contraception.2011.07.013. Epub 2011 Aug 24. PMID 22018121
- [Background] Conde-Agudelo A, Rosas-Bermudez A, Kafury-Goeta AC. Effects of birth spacing on maternal health: a systematic review. Am J Obstet Gynecol. 2007 Apr;196(4):297-308. doi: 10.1016/j.ajog.2006.05.055. PMID 17403398
- [Background] Thiel de Bocanegra H, Chang R, Howell M, Darney P. Interpregnancy intervals: impact of postpartum contraceptive effectiveness and coverage. Am J Obstet Gynecol. 2014 Apr;210(4):311.e1-311.e8. doi: 10.1016/j.ajog.2013.12.020. Epub 2013 Dec 13. PMID 24334205
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] Rose SB, Lawton BA. Impact of long-acting reversible contraception on return for repeat abortion. Am J Obstet Gynecol. 2012 Jan;206(1):37.e1-6. doi: 10.1016/j.ajog.2011.06.102. Epub 2011 Jul 13. PMID 21944222
- [Background] Madden T, Mullersman JL, Omvig KJ, Secura GM, Peipert JF. Structured contraceptive counseling provided by the Contraceptive CHOICE Project. Contraception. 2013 Aug;88(2):243-9. doi: 10.1016/j.contraception.2012.07.015. Epub 2012 Sep 5. PMID 22959396
- [Background] Peipert JF, Zhao Q, Allsworth JE, Petrosky E, Madden T, Eisenberg D, Secura G. Continuation and satisfaction of reversible contraception. Obstet Gynecol. 2011 May;117(5):1105-1113. doi: 10.1097/AOG.0b013e31821188ad. PMID 21508749
- [Background] Finer LB, Jerman J, Kavanaugh ML. Changes in use of long-acting contraceptive methods in the United States, 2007-2009. Fertil Steril. 2012 Oct;98(4):893-7. doi: 10.1016/j.fertnstert.2012.06.027. Epub 2012 Jul 13. PMID 22795639
- [Background] Randel A. Guidelines for the use of long-acting reversible contraceptives. Am Fam Physician. 2012 Feb 15;85(4):403-4. No abstract available. PMID 22335322
- [Background] Zuckerman B, Nathan S, Mate K. Preventing unintended pregnancy: a pediatric opportunity. Pediatrics. 2014 Feb;133(2):181-3. doi: 10.1542/peds.2013-1147. Epub 2014 Jan 27. No abstract available. PMID 24470643
- [Background] American Academy of Pediatrics Committee on Adolescence: Contraception and adolescents. Pediatrics. 1990 Jul;86(1):134-8. No abstract available. PMID 2359670
- [Background] Jones J, Mosher W, Daniels K. Current contraceptive use in the United States, 2006-2010, and changes in patterns of use since 1995. Natl Health Stat Report. 2012 Oct 18;(60):1-25. PMID 24988814
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Cwiak C, Gellasch T, Zieman M. Peripartum contraceptive attitudes and practices. Contraception. 2004 Nov;70(5):383-6. doi: 10.1016/j.contraception.2004.05.010. PMID 15504377
- [Background] Hladky KJ, Allsworth JE, Madden T, Secura GM, Peipert JF. Women's knowledge about intrauterine contraception. Obstet Gynecol. 2011 Jan;117(1):48-54. doi: 10.1097/AOG.0b013e318202b4c9. PMID 21173643